CLINICAL TRIAL: NCT05633849
Title: Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Pro Resolve® Sports on Treatment of Patients With Symptomatic Knee Osteoarthritis
Brief Title: Evaluation of the Effect of Pro Resolve® Sports on Treatment of Patients With Symptomatic Knee Osteoarthritis
Acronym: GAUDÍ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Solutex GC S.L. (Industry)
Collaborators: OAFI Foundation (Osteoarthritis Foundation International) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GAUDÍ
Record Dates: First submitted 2022-10-31; First posted 2022-12-01 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Knee Osteoarthritis
Keywords: SPMs; Resolvins; Osteoarthritis; Pain; Quality of life
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain

STUDY DESIGN:
Intervention Model Description: randomized, multicentre, double-blind, placebo-controlled, parallel-group pilot study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): In placebo group, participants were instructed to take two 500 mg olive oil placebo (placebo group) after breakfast and two after dinner during the first 6 weeks of the study. During the next 6 weeks, participants were instructed to take one softgel after breakfast and one after dinner. Thus, the treatment period was 12 weeks
  Interventions: Dietary Supplement: Placebo group
- Specialized pro-resolving mediators (SMP) group (Experimental): In SPM group, Participants were instructed to take two 500 mg softgels of LIPINOVA after breakfast and two after dinner during the first 6 weeks of the study. During the next 6 weeks, participants were instructed to take one softgel after breakfast and one after dinner. Thus, the treatment period was 12 weeks
  Interventions: Dietary Supplement: SMP group

INTERVENTIONS:
Dietary Supplement: SMP group — Participants were instructed to take two 500 mg softgels of LIPINOVA(SPM group) after breakfast and two after dinner during the first 6 weeks of the study. During the next 6 weeks, participants were instructed to take one softgel after breakfast and one after dinner. Thus, the treatment period was 12 weeks
  Arms: Specialized pro-resolving mediators (SMP) group
Dietary Supplement: Placebo group — Participants were instructed to take two 500 mg softgels of olive oil placebo after breakfast and two after dinner during the first 6 weeks of the study. During the next 6 weeks, participants were instructed to take one softgel after breakfast and one after dinner. Thus, the treatment period was 12 weeks
  Arms: Placebo group

SUMMARY:
The GAUDI study was a randomized, multicentre, double-blind, placebo-controlled, parallel-group pilot study conducted in 5 Spanish sites.

Eligible patients were adults younger than 68 years diagnosed with symptomatic knee Osteoarthritis and pain score (VAS) ≥ 5.

The primary endpoint was the change in pain from baseline to week 12. Secondary endpoints included the comparison in the change of pain, stiffness, and function according to the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) between groups from baseline to week 12, the assessment of the constant, intermittent, and total pain according to OMERACT-OARSI score, the changes in health-related quality of life score measured by the EUROQoL-5 questionnaire (16) between both study groups, the use of rescue, and anti-inflammatory medication, and the incidence of adverse events (AEs) during the study.

DETAILED DESCRIPTION:
The GAUDI study was a randomized, multicentre, double-blind, placebo-controlled, parallel-group pilot study conducted in 5 Spanish centers in compliance with the World Medical Association Declaration of Helsinki, all its amendments, and national regulations. The Independent Ethic Committee of Hospital U. La Paz (Madrid, Spain) approved this study. All patients gave their written informed consent.

The study duration was 24 weeks, including a screening period, a treatment period with monthly visits from the start of the study until week 12, and a follow-up visit 24 weeks after the study initiation conducted by telephone call.

Participants were instructed to take two 500 mg softgels of LIPINOVA(SPM group) or olive oil placebo (placebo group) after breakfast and two after dinner during the first 6 weeks of the study. During the next 6 weeks, participants were instructed to take one softgel after breakfast and one after dinner. Thus, the treatment period was 12 weeks.

Eligible patients were adults younger than 68 years diagnosed with symptomatic knee OA (according to the American College of Rheumatology [ACR]), primary knee (OA), confirmed 2-3 Kellgren and Lawrence radiologic degree (15), and pain Visual Analogue Scale (VAS) score ≥ 5. Patients were excluded if they were allergic to fish or seafood, had an arthroscopy within the last year, had been diagnosed with secondary knee osteoarthritis, cardiopathy, pneumopathy, non-compensated nephropathy, neuropathy affecting mobility, non-compensated psychiatric disorder, fibromyalgia, and/or cognitive disorder. Patients were also excluded if they had received chondroitin sulfate, glucosamine, diacerein, corticoids infiltration, and/or platelet-rich plasma infiltration in the knee three months before the study inclusion, NSAIDs three weeks before the inclusion, and/or hyaluronic acid infiltration in the knee six months before the inclusion. Patients could not have had a drug abuse record three years before the inclusion and have participated in another clinical trial.

The primary endpoint was the change in pain measured on a VAS from baseline to week 12. Secondary endpoints included the comparison in the change of pain, stiffness, and function according to the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) between groups from baseline to week 12, the assessment of the constant, intermittent, and total pain according to OMERACT-OARSI score, the changes in health-related quality of life score measured by the EUROQoL-5 questionnaire (16) between both study groups, the use of concomitant, rescue, and anti-inflammatory medication, and the incidence of adverse events (AEs) during the study.

ELIGIBILITY:
Inclusion Criteria:

* Adults younger than 68 years
* Diagnosis of symptomatic knee OA (according to the American College of Rheumatology [ACR]), primary knee (OA)
* Patients with primary knee arthrosis
* Patients with confirmed 2-3 Kellgren and Lawrence radiologic degree
* Patients with pain Visual Analogue Scale (VAS) score ≥ 5
* Patients that signed informed consent

Exclusion Criteria:

* Patients allergic to fish or seafood
* Patients that had an arthroscopy within the last year
* Patients that had been diagnosed with secondary knee osteoarthritis
* Patients with concomitant illnesses such as cardiopathy, pneumopathy, non-compensated nephropathy, neuropathy affecting mobility, non-compensated psychiatric disorder, fibromyalgia, and/or cognitive disorder
* Patients that have received NSAIDs during last 3 weeks previous to join the study
* Patients that hace received chondroitin sulfate, glucosamine, diacerein, corticoids infiltration, and/or platelet-rich plasma infiltration in the knee three months before the study inclusion
* Patients that have had a drug abuse record three years before the inclusion
* Patients that have had a drug abuse record three years before the inclusion

Ages: 18 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2021-10-14 (Actual); Study Completion 2021-10-14 (Actual)

PRIMARY OUTCOMES:
Change in Pain | Basal and 12 weeks
  Change in pain measured on a visual analogic scale (VAS) (intragroup). Min: 0 (no pain) max: 10 (the worst pain possible)

SECONDARY OUTCOMES:
Change in Pain (between groups) assessed by Visual Analogic Scale. Min: 0 (no pain) max: 10 (the worst pain possible) | Basal and 12 weeks
  Change in pain (between groups)
Use of Rescue medication and patient drop-outs | Basal and 12 weeks
  Percentage of patients that drops-out the study and percentage of patients that need to use rescue medication during the study
Change in functionality assessed by WOMAC (Eastern Ontario McMaster Universities Osteoarthritis Index) score | Basal and 12 weeks
  Changes in functionality using WOMAC score. Min: 0 (better), max: 96 (worse)
Safety of study product, assessed as percentage of patients suffering adverse events related to study product | 12 weeks
  % of adverse events related to study product
Changes in pain assessed as changes in OMERACT-OARSI score | Basal and 12 weeks
  Changes in OMERACT-OARSI score. Min: 0 (better), max 44 (worse)
Quality of life of patients assessed as changes in EQ-5D-5L score | Basal and 12 weeks
  Changes in Quality of life (EQ-5D). Visual analogue scale (quantitative): min: 0 (worse), max: 100 (better). qualitative variables: mobility, self-care, usual activities, pain/discomfort, anxiety/depression Min: 1 (better); max: 5 (worse)
Inflammatory biomarkers: C-reactive protein (CRP) | Basal and 12 weeks
  Changes in Inflammatory biomarkers: CRP
Inflammatory biomarkers: Interleukin -1 (IL-1) | Basal and 12 weeks
  Changes in Inflammatory biomarkers: IL-1
Inflammatory biomarkers: Interleukin-6 (IL-6), | Basal and 12 weeks
  Changes in Inflammatory biomarkers: IL-6
Inflammatory biomarkers: Interleukin-8 (IL-8) | Basal and 12 weeks
  Changes in Inflammatory biomarkers: IL-8
Inflammatory biomarkers: Tumoral Necrosis Factor -α (TNF-α) | Basal and 12 weeks
  Changes in Inflammatory biomarkers: TNF-α

CONTACTS AND LOCATIONS:
Overall Officials: Gil Rodas, MD, Principal Investigator — Medical Services F.C. Barcelona
Locations (5):
- Spain (5):
  - Clínica Segura, Las Rozas de Madrid, Madrid
  - Clínica Dr. Rodas, Avilés, Principality of Asturias
  - Medical Services Ath, Club Bilbao, Bilbao, Vizcaya
  - Instituto Poal de Reumatología, Barcelona
  - Medical Services F.C. Barcelona, Barcelona

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moller I, Rodas G, Villalon JM, Rodas JA, Angulo F, Martinez N, Verges J. Randomized, double-blind, placebo-controlled study to evaluate the effect of treatment with an SPMs-enriched oil on chronic pain and inflammation, functionality, and quality of life in patients with symptomatic knee osteoarthritis: GAUDI study. J Transl Med. 2023 Jun 29;21(1):423. doi: 10.1186/s12967-023-04283-4. PMID 37386594